CLINICAL TRIAL: NCT06564207
Title: Randomized, Double-Blinded, Placebo-Controlled Phase 2 Study for the Long Term Evaluation of Fostamatinib for the Treatment of Adult Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Fostamatinib for Treating Acute Respiratory Distress Syndrome (ARDS) in Hospitalized Adults
Acronym: FOSTA-ARDS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Rigel Pharmaceuticals (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INOVA-2023-169
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — fostamatinib

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to receive either fostamatinib plus standard of care or placebo plus standard of care.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) + Placebo (BID for 14 Days) (Placebo Comparator): Participants randomized to this arm will receive standard of care (SOC) treatment plus placebo given twice daily for 14 days
  Interventions: Drug: Placebo
- Standard of Care (SOC) + Fostamatinib 150mg (BID for 14 Days) (Experimental): Participants randomized to this arm will receive standard of care (SOC) treatment plus fostamatinib 150mg given twice daily for 14 days
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Placebo — Placebo to be given twice daily for 14 days
  Arms: Standard of Care (SOC) + Placebo (BID for 14 Days)
Drug: Fostamatinib — Fostamatinib 150mg to be given twice daily for 14 days
  Other Names: fostamatinib disodium
  Arms: Standard of Care (SOC) + Fostamatinib 150mg (BID for 14 Days)

SUMMARY:
This study is designed to evaluate the safety and efficacy of fostamatinib in hospitalized adult participants with acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase 2 study for long-term evaluation of fostamatinib for the treatment of adult patients with acute respiratory distress syndrome. Subjects will be randomly assigned 1:1 to either standard of care treatment plus fostamatinib or standard or care plus placebo. Th study drug will be taken twice daily for 14 days.

The primary objective will be to evaluate drug safety in hospitalized patients with severe ARDS. Other objectives include assessment of the efficacy and clinically relevant endpoints, such as mortality and effects on resolution of this disease entity. The ability of fostamatinib to impact the short term and long term outcomes for patients with ARDS will be directly evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Subject (or legal representative) provides informed consent to study participation.
* Subject (or legal representative) understands and agrees to comply with planned study procedures.
* Hospitalized with acute respiratory failure from ARDS with ratio of partial pressure of arterial oxygen to fraction of inspired oxygen PaO2/FiO2 of 200 mm of Hg or less with positive end expiratory pressure (PEEP) equal to or higher than 5 cm of H2O and requiring invasive mechanical ventilation or extracorporeal support.
* Functional respiratory imaging (FRI) compatible CT scan of the chest within the prior 7 days.
* Duration of invasive mechanical ventilation < 10 days.
* Females of childbearing potential must agree to be abstinent or seek a highly effective form of contraception from the time of enrollment through 30 days after the last day of study drug.

Exclusion Criteria:

* Severe hepatic impairment (Child-Pugh Class C).
* Abnormal liver function tests (AST or ALT > 3x ULN or AST or ALT > 3x ULN)
* Pregnant or nursing.
* Participation in any other clinical trial, or receipt of an investigational medicinal product within 30 days prior.
* Known concomitant life-threatening disease with a life expectancy < 6 months.
* Known hypersensitivity to fostamatinib.
* Uncontrolled hypertension (Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg).
* Neutrophil count < 1000/uL
* Death expected within 72 hours
* Received a live vaccine in the last 30 days
* Those who were cognitively impaired or mentally disabled prior to acute illness
* Patients with acute coronary syndrome, ejection fraction <30%, or active unstable arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-08-30 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Incidence of Serious Adverse Events (SAEs) Through Day 30 | Up to 30 days post-intervention
  The cumulative incidence of serious adverse events (SAEs) occurring through day 30 following the intervention. An SAE is defined by the International Conference on Harmonization (ICH) guidelines as any adverse event fulfilling at least one of the following criteria:
  Results in death; Is life threatening; Requires in-subject hospitalization or prolongation of an existing hospitalization; Results in persistent or significant disability/incapacity; Is considered an important medical event (or medically significant)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S. King, MD, FACP, Principal Investigator — Inova Schar Heart and Vascular

IPD SHARING:
Plan to Share IPD: No